CLINICAL TRIAL: NCT01665534
Title: Procalcitonin and the Inflammatory Response to Salt in Essential Hypertension: a Randomised Cross-over Clinical Trial.
Brief Title: Inflammatory Response to Salt in Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carmine Zoccali (Other Government)
Responsible Party: Sponsor-Investigator, Carmine Zoccali, Director of the Nephrology, Dialysis and Transplantation Unit and Project Leader of the Section of "Clinical Epidemiology and Pathophysiology of Renal Diseases and Hypertension" of CNR-IBIM, Reggio Calabria, Italy, Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy
Organization: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SS-011-RC
Record Dates: First submitted 2012-08-07; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Essential Hypertension.
Keywords: hypertension; inflammation; salt intake
MeSH Terms: conditions — Essential Hypertension; Hypertension; Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Effect of salt intake (Experimental): During the high salt intake period, patients received a 10-20 mmol sodium diet plus sodium tablets (180 mEq/die) to achieve a 200 mmol intake /day for two weeks. During the low salt intake period, patients received a 10-20 mmol sodium diet + placebo tablets for two weeks.
  Interventions: Behavioral: High salt intake

INTERVENTIONS:
Behavioral: High salt intake — During the high salt intake period, patients received a 10-20 mmol sodium diet plus sodium tablets (180 mEq/die) to achieve a 200 mmol intake /day for two weeks

SUMMARY:
Salt is a main environmental risk factor involved in atherosclerotic complications and in the high risk of a variety of cardiovascular (CV) diseases including hypertension, left ventricular hypertrophy (LVH), chronic kidney disease (CKD) and heart failure. The link between sodium and cardiovascular disease is complex and involves blood pressure (BP) dependent and independent mechanisms. Among the latter, inflammation is suspected to be a major effector of arterial damage brought about by the salt excess in animal models. In humans, C-Reactive Protein (CRP) associated directly with dietary salt intake in a population-based survey but such a link was not confirmed in other studies. This apparent discrepancy may depend on the observational (i.e., open to confounding) nature of these studies. Inflammatory cytokines are essential for the short term systemic response to environmental stressors. For example it is well established that TNF-α, a cytokine that modulates renin gene expression by signalling via TNF-receptor 2, exerts a protective effect for the myocardium in a stressful condition like experimental cardiac ischemia while low levels of adiponectin have a detrimental effect in the same setting. Thus, the inflammation-sodium relationship may be non-linear and severe salt restriction may actually trigger inflammation, a hypothesis suggested by the observation that biomarkers of inflammation rose in response to salt depletion in a sequential study in essential hypertensives. However, the lack of randomization in this study leaves open the question whether the observed pro-inflammatory effect was due to change in salt intake or to other, unmeasured time-dependent effect(s). With this background in mind the investigators setup a randomized, single masked, cross-over study to assess the effect of a short term very low salt diet on biomarkers of innate immunity in patients with uncomplicated essential hypertension.

DETAILED DESCRIPTION:
The protocol was in conformity with the ethical guidelines of our institution and informed consent was obtained by each participant. During the run-in phase of the study, which lasted 1 month, patients underwent standard arterial pressure measurements on two separate occasions (at least 10 days apart) and were considered eligible for the study if their casual arterial pressure exceeded 140/90 mmHg.

Patients were randomized to either a 10-20 mmol sodium diet plus sodium tablets (180 mEq/die) to achieve a 200 mmol intake /day, or the same diet plus identical placebo tablets, each for two weeks. At the end of each of these two-week periods, all patients underwent a 24-hours urine collection, a fasting blood sampling and a 24h ambulatory blood pressure monitoring (see below).

Ambulatory monitoring was performed with a device conforming with the AAMI criteria (Takeda 2420 model 7, Takeda Medical, Osaka, Japan). Between 08.30 and 11.30 hours, after placement of the device in the left (non-dominant) arm, the patients rested quietly in an armchair for 15 min and arterial pressure was taken automatically three times (at 5 min intervals). Patients then went home and remained indoors throughout all the recording day. They were instructed to spend a relaxed, quiet day avoiding physical efforts. Recordings were set at 15 min intervals between the 07.00 to 22.00 hours and every 30 min during the sleeping hours (22.00 pm to 07.00). The calibration of the ambulatory recorder was performed against a mercury sphygmomanometer before each recording. Patients were classified as salt-sensitive if the changes in mean arterial pressure between low and high salt diet was > 10%.

Blood sampling was performed on the last day of each period after 45 minutes supine rest. The patients were specifically instructed not to alter their smoking habits, alcohol and coffee intake and not to modify the level of physical activity throughout the study.

Urinary sodium was measured by an ion-selective electrode using a Beckman (Fullertone, CA, USA) EA-2 Electrolyte Analyser. Serum and urine creatinine was measured by a colorimetric method using a COBAS-Mira spectrophotometer (Roche, Basel, Switzerland). The measurements of plasma renin activity (PRA) and plasma aldosterone concentration were performed by radioimmunoassay (RIA) using a commercially available kit (Technogenetics-Milan, Italy).

Biomarkers of inflammation and endothelial integrity/function High sensitivity C-Reactive Protein (hs-CRP) was measured in plasma by a nephelometric method (Dade-Behring, Scoppito, L'Aquila, Italy) (intra-assay CV: 3.5%; inter-assay CV: 3.4%; normal range < 2.87 mg/L). Interleukin-6 (intra-assay CV: 2.6%; inter-assay CV: 4.5%, normal range < 12.5 pg/mL) and TNF-α (intra-assay CV: 4.7%; inter-assay CV: 5.8%, normal range < 15.6 pg/mL) were measured by commercially available RIA kits (R&D System, Minneapolis, USA). High sensitivity procalcitonin (PCT) (intra-assay CV: 2-3% normal value < 0.05 ng/mL) was measured by an immunofluorescence method (Kriptor, BRAHMS, Henningsdorf, Germany). Plasma Adiponectin (intra-assay CV: 3.9%; inter-assay CV: 8.4%) and Leptin (intra-assay CV: 5.0%; inter-assay CV: 4.5%) were measured by a RIA kit (Linco Research Missouri, USA).

ELIGIBILITY:
Inclusion Criteria:

Patients with uncomplicated, untreated essential hypertension (age>18 years).

Exclusion Criteria:

Patients with secondary hypertension, liver disease, neoplasia and other chronic disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline of inflammatory biomarkers (TNF-alpha, procalcitonin, IL-6, C-Reactive Protein, adiponectin and leptin) in response to salt intake. | Inflammatory biomarkers were measured at baseline and at the end of two-week diet periods.
  Patients were randomized to either a 10-20 mmol sodium diet plus sodium tablets (180 mEq/die) to achieve a 200 mmol intake /day, or the same diet plus identical placebo tablets, each for two weeks.

SECONDARY OUTCOMES:
Blood pressure response to salt intake. | 24h ambulatory blood pressure was measured at baseline and at the end of two-week diet periods.
  Patients were randomized to either a 10-20 mmol sodium diet plus sodium tablets (180 mEq/die) to achieve a 200 mmol intake /day, or the same diet plus identical placebo tablets, each for two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Zoccali, Prof., Study Chair — Nephrology, Dialysis and Transplantation Unit and CNR-IBIM